CLINICAL TRIAL: NCT05764811
Title: Mechanism of the Effect by Sodium-glucose Cotransporter-2 Inhibitor on Obesity Associated Cardiomyopathy
Brief Title: SGLT-2 Inhibitor Effects on Cardiac and Hepatic Metabolic Profiles for the Diabetes Patients Combined With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ping-Yen Liu, Doctor/Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-BR-108-103
Record Dates: First submitted 2023-01-26; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Fatty Liver Disease
Keywords: fatty liver; diabetes mellitus; SGLT2 inhibitor
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Diabetes Mellitus | interventions — Canagliflozin; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canagliflozin Treatment (Active Comparator): Use Canagliflozin 100 mg daily, 1 month
  Interventions: Drug: Canagliflozin 100mg
- non-Canagliflozin Treatment (No Intervention): Standard treatment

INTERVENTIONS:
Drug: Canagliflozin 100mg — 100 mg daily for a month
  Other Names: standard of care
  Arms: Canagliflozin Treatment

SUMMARY:
Obesity is closely associated with an increased risk of cardiomyopathy because of the high metabolic activity of excessive fat while effective treatment of obesity-related cardiomyopathy is currently unsolved. Sodium-glucose cotransporter-2 inhibitors (SGLT2-i) are a class of diabetic medications. Besides improving glucose control, SGLT2-i has been shown to be able to reduce the bodyweight as well as the mortality and hospitalization rates for heart failure and cardiovascular disease in the type 2 diabetes patients. It has been proposed that the heart protection by SGLT2-i might be caused by modulating the production of adipokine and cytokine. The investigators will enrolled 40 patients (diabetes mellitus with BMI>27 Kg/m2) from obesity weight-reduction clinics: 1) 20 patients treated with SGLT2-i (CANA) and regular weight-reduction plan; 2) 20 patients with regular weight reduction plan, without CANA, for 4 weeks. The investigators will compare the variation of Fibroblast growth factor-21 (FGF21) related proteins and RNA between these 2 groups of subjects. The investigators will arrange cardiac ultrasound, hepatic MRI and fibroscan, body composition dual energy x-ray absorptiometry to evaluate the possible mechanisms underlying the liver and heart modification process, as a scientific basis for precision medicine in the future. Conclusions: SGLT2-i treatment may increase the concentration of FGF21, either in the liver or heart, thus to protect the high-fat diet induced obesity associated heart dysfunction by activating FGF21 downstream protein expression.

DETAILED DESCRIPTION:
The investigators will enrolled 40 diabetes mellitus with BMI>27 Kg/m2 patients from obesity weight-reduction clinics and will compare the variation of FGF21 related proteins between these 2 groups of subjects. Serial examinations will evaluate the possible mechanisms underlying the protective mechanism. This investigation expect that SGLT2-inhibitor can increase the concentration of FGF21 in the heart by increasing FGF21 in the liver, thereby modifying associated protein expressions and ultimately improving cardiac function and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 20 years of age
2. With diagnosis of diabetic mellitus (HbA1C≧6.5%) by medical record or physicians
3. BMI ≧ 27 kg/m2, which is the current definition of obesity from Health Promotion Administration, Ministry of Health and Welfare.

Exclusion Criteria:

1. Unwilling to participating current clinical trial
2. Cannot tolerate SGLT2-i therapy
3. Not willing to join the study
4. History of failure treatment experience from SGLT2-i or other weight reduction plan
5. Received pharmaceutical or clinical trials within past 1 year

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
measure the severity of fatty liver via MRI | 4 weeks
  The fibrotic score and severity by MRI of the liver will be performed before and after the treatment. The measurement of fatty liver requires both in-phase (IP) and out-of-phase (OOP) imaging to be adequately assessed. Fatty liver appears: T1: hyperintense, T2: mildly hyperintense, IP/OOP imaging: signal drop out on OOP imaging On IP/OOP imaging, signal loss is demonstrated when there is 10-15% fat fraction with maximum signal loss occurring when there is 50% fatty infiltration of the liver. In situations in which there is >50% fatty infiltration, the out-of-phase sequence paradoxically becomes less hypointense than at 50%.

SECONDARY OUTCOMES:
measure the body weight before and after the treatment | 4 weeks
  check the status of body weight (kilograms) before and after treatment
measure the body height before and after the treatment | 4 weeks
  check the status of body height (metres) before and after treatment
measure the body mass index (BMI) before and after the treatment | 4 weeks
  compare BMI before and after treatment; BMI is a value derived from the mass (weight) and height of a person. The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m2, resulting from mass in kilograms and height in metres.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Yen Liu, Study Director — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No